CLINICAL TRIAL: NCT00569296
Title: A Phase I Study of Anti-CD3 x Cetuximab-Armed Activated T Cells, Low Dose IL-2, and GM-CSF for EGFR-Positive, Advanced Non-Small Cell Lung Cancer
Brief Title: Laboratory-Treated Autologous Lymphocytes, Aldesleukin, and GM-CSF in Treating Patients With Recurrent, Refractory, or Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000577502; 349-32 (Other: Roger Williams Medical Center); 3422 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — aldesleukin; Interleukin-2; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T-cells (Experimental): EGFRBi-armed autologous activated T cells
  Interventions: Biological: EGFRBi-armed autologous activated T cells; Biological: aldesleukin; Biological: sargramostim

INTERVENTIONS:
Biological: EGFRBi-armed autologous activated T cells — Dose escalation, dosage depends on when entered in study. 8 infusions (twice a week over 4 weeks. Each infusion will be over at least 1 hour.
Biological: aldesleukin — 300,00IU/m2/day beginning 3 days before the first Activated T-cell infusion and ending 1 week after the last infusion
  Other Names: IL-2
Biological: sargramostim — 250 micrograms/m2/twice weekly beginning 3 days before the first activated T-cell infusion and ending 1 week after the last Activated T-cell infusion
  Other Names: GM-CSF

SUMMARY:
RATIONALE: Giving autologous lymphocytes that have been treated in the laboratory with antibodies may stimulate the immune system to kill tumor cells. Aldesleukin may stimulate the lymphocytes to kill tumor cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving laboratory-treated autologous lymphocytes together with aldesleukin and GM-CSF may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of laboratory-treated autologous lymphocytes when given together with aldesleukin and GM-CSF in treating patients with recurrent, refractory, or metastatic non-small cell lung cancer.

FUNDING SOURCE--FDA OOPD

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and maximum tolerated dose of EGFRBi-armed autologous activated T-cells (ATC) when administered in combination with low-dose aldesleukin and sargramostim (GM-CSF) in patients with recurrent, refractory, or extensive (metastatic) non-small cell lung cancer (NSCLC).

Secondary

* Assess clinical outcome based on tumor responses, overall survival, and progression-free survival.
* Monitor changes in sera concentrations of the tumor marker in association with EGFRBi-armed ATC administration throughout the study and at time points thereafter in patients with elevated levels of carcinoembryonic antigen (CEA) prior to beginning the study.
* Monitor patient sera for human anti-mouse antibodies (HAMA).
* Evaluate immune response, which may reflect immune augmentation in response to EGFRBi-armed ATC infusions, in peripheral blood mononuclear cell (PBMC) samples as well as purified immune cell populations.
* Investigate proliferation in response to ex vivo stimulation with NSCLC tumor-associated antigens, sera cytokine profiles (Th1 vs Th2), cytotoxicity of patient PBMC, and interferon gamma ELISPOTS as a surrogate marker for assessing generation of EGFR-specific cytotoxic T-lymphocytes (CTL).

OUTLINE: Peripheral blood mononuclear cells (PBMCs) are collected by 1 or 2 leukaphereses for the generation of activated T cells (ATCs). The PBMCs are activated with OKT3 (anti-CD3) and expanded in aldesleukin for up to 14 days. The ATCs are then armed with EGFRBi.

Patients receive EGFRBi-armed autologous ATCs IV over 30-60 minutes twice weekly for 4 weeks (a total of 8 infusions) in the absence of disease progression or unacceptable toxicity. Patients also receive low-dose aldesleukin subcutaneously (SC) once daily and sargramostim (GM-CSF) SC twice weekly beginning 3 days before the first ATC infusion and continuing for 1 week after the last ATC infusion.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Recurrent, refractory, or metastatic disease after ≥ 1 prior first-line regimen (chemotherapy or radiotherapy)
* Documented EGFR-positive disease (any expression level) by immunohistochemistry (IHC) (may be based on archival sample)
* Measurable or evaluable disease by radiograph, CT scan, MRI, and/or physical exam
* Appropriate slides of the primary lesion must be available for review of IHC staining assessment by a central pathology team
* No clinical evidence of active brain metastases

  * Patients with brain metastases are eligible provide they have received definitive radiotherapy or chemotherapy and/or have undergone surgical resection for brain metastases
* No prior hematological malignancy

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 60-100% OR ECOG PS 0-2
* Life expectancy ≥ 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Granulocytes ≥ 1,000/mm^3
* Platelet count ≥ 50,000/mm^3
* Hemoglobin ≥ 8 g/dL
* BUN ≤ 2.0 times normal
* Serum creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 1.5 times normal
* SGOT ≤ 1.5 times normal (with or without liver metastases)
* Hepatitis B surface antigen and HIV negative
* LVEF ≥ 45 % at rest (by MUGA)

  * No evidence of depressed left ventricular function
* FEV_1, DLCO, and FVC ≥ 50% of the predicted value
* No other malignancy, except for the following:

  * History of curatively treated in situ squamous cell carcinoma or basal cell carcinoma of the skin
  * History of other curatively treated malignancy (except those with a hematologic origin) for which the patient has remained in complete remission > 5 years after completing therapy (as documented by history, physical exams, tumor markers, and radiology scanning)
* No serious medical or psychiatric illness that would preclude giving informed consent or receiving intensive treatment
* No recent myocardial infarction (within the past year)
* No current angina/coronary symptoms requiring medications
* No clinical evidence of congestive heart failure requiring medical management (irrespective of MUGA results)
* No systolic blood pressure (BP) ≥ 130 mm Hg or diastolic BP ≥ 80 mm Hg

  * Patients with elevated BP must have it controlled by anti-hypertensive medications for at least 7 days prior to the first infusion

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy or radiotherapy
* At least 4 weeks since prior cetuximab or small molecule EGFR-inhibitors including, but not limited to, gefitinib or erlotinib hydrochloride
* No concurrent radiotherapy
* No concurrent steroids except for treatment of adrenal failure, septic shock, or pulmonary toxicity or hormones for non-disease-related conditions (e.g., insulin for diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety | 4 weeks
Maximum tolerated dose of EGFRBi-armed autologous activated T-cells | 4 weeks
Determination of immunologic changes by evaluation of cytokine profiles obtained before and after stimulation with OKT3 in vitro | 4 weeks

SECONDARY OUTCOMES:
Overall survival | 2 years
Progression-free survival | 2 years
Evaluation of tumor markers and human anti-mouse antibody responses as assessed by carcinoembryonic antigen (CEA) levels in serum samples and development of IgG and IgM anti-mouse antibody responses to the Bi-antibodies | 4 weeks
Determination of immunologic changes by evaluation of peripheral blood lymphocytes | 4 weeks
Determination of immunologic changes by evaluation of cytotoxic T-lymphocytes as measured by interferon gamma ELISPOTS directed at autologous tumor or lung cancer cell lines | 4 weeks
Determination of immunologic changes by evaluation of phenotypes of peripheral blood mononuclear cells before and after immunotherapy | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Abby Maizel, MD, PhD, Study Chair — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States